CLINICAL TRIAL: NCT04447742
Title: Bern Birth Cohort / Trajectory of Microbiota Maturation in Healthy Bern Infants - a Network Approach
Acronym: BeBiCo
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-00510; 3962 (Other: Direktion Lehre und Forschung Insel Spital Bern)
Record Dates: First submitted 2020-05-19; First posted 2020-06-25 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Maturation of the Healthy Infant Intestinal Microbiota; Microbial Colonization; Nutrition Disorder, Infant; Milk Expression, Breast; Mental Health Disorder
MeSH Terms: conditions — Communicable Diseases; Infant Nutrition Disorders; Breast Milk Expression; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Maternal stool samples
  * Maternal milk samples
  * Maternal skin swabs
  * Maternal vaginal swabs (optional)
  * Infant stool samples infant skin swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Intestinal microbiota composition is fundamental to human health and undergoes critical changes within the first two years of life. Factors probably influencing the microbiota are the maternal microbiota and the general environment in Switzerland. However, the development of the intestinal microbiota is incompletely understood. Gaining knowledge of the trajectory of microbiota maturation is likely key to the understanding of the pathogenesis of many pathologies in childhood.

Aims: The investigators aim for a deep understanding of the maturation of the healthy infant intestinal microbiota regarding composition, diversity and metabolic activities. The investigators aim for identifying parameters affecting microbiota maturation and effects of the microbiota on infant outcome.

Methods: The investigators will recruit 250 pregnant mothers who will be followed as mother-baby pairs until 10 years of age. Infants will be followed clinically to determine adequate growth and development as well as pathology including abdominal pain. Epidemiological parameter and infant nutrition will be assessed. The investigators will collect biological samples such as stool, maternal milk, vaginal swaps and skin swaps.

Species composition and diversity will be assessed by 16S sequencing. Metagenomic shotgun sequencing and bacterial messenger ribonucleic acid (mRNA) analysis will inform about metabolic potential and metabolic activity of the microbiota. Mass spectrometry will assess the small molecule content of stool and maternal milk samples. Network analysis will be used to assess the complex relationships between bacteria metabolic activities and small molecular content.

Expected results: The investigators expect an increase in complexity and metabolic potential and activity with age. Microbiota parameters will differ according to nutrition and might predict infant outcomes such as growth and abdominal pain. Systematic analysis of sequential maternal and infant bacteria samples from stool, skin and maternal milk will help characterizing bacterial transfer from mother to infant Conclusion: The investigators propose an observational study of healthy Bern mother baby pairs with clinical characterisation and biological sampling. Advanced analysis tools will be used to characterise the microbiota and address mechanistic questions.

DETAILED DESCRIPTION:
Methods for sample analysis:

For the primary objective and outcome/ endpoint of the study, bacterial content of infant stool will be analyzed by:

* Mass spectrometry to assess intestinal content (metabolome). Techniques have been established in the laboratory of Prof. U. Sauer who already collaborated with the investigators' group in previous studies.
* 16S ribosomal ribonucleic acid (rRNA) sequencing for bacterial species composition as well as microbial diversity.
* Bacterial full genome metagenomics shotgun sequencing to identify bacterial genes present (metabolic potential of the microbiota).
* Bacterial mRNA sequencing to assess transcription and a functional role of the microbiota (metabolic activity of microbiota).
* Analysis of the intestinal virome and eukaryotic intestinal populations by appropriate sequencing or culturing techniques.
* Analysis of IgA antibodies in human milk and stool and the interaction of antibodies with intestinal bacteria.

For the secondary endpoints identical analyses will be performed in skin swabs, maternal milk, maternal vaginal swabs and maternal stool. Parameters for infant growth, neurodevelopment, immune maturation and potential occurrence of pathology will be assessed at every visit. Maternal and infant nutrition, hygiene, socioeconomic status and clinical history will be assessed by questionnaires at every visit. Milk samples will further be analyzed for their cellular contents by flow cytometry and single cell RNA-sequencing, as well as for cytokines and exosome-based miRNAs. All biosamples will be analyzed by mass spectrometry to assess impact of the environment on infant metabolism and physiology.

Further follow-up experiments with the acquired samples are possible. Specifically, individual bacteria strains can be isolated and cultured in vitro and also tested alone or in combination in experimental animals.

Bacterial sequencing by the methods described above will also inevitably identify maternal or infant DNA sequences, since metagenomic shotgun sequencing cannot differentiate between bacterial and human DNA. These human DNA sequences will not be analyzed within the scope of this project. However, these sequences might be the subject of future studies. Study participants will therefore be asked for permission to analyze human DNA from mother and/ or child at the page for "further analyses" within the consent form. An option to "opt out" for human DNA analysis will be provided and refusal will not lead to exclusion from the study.

Any findings of clear relevance to the health of the participant (i.e. mother or child) will be reported to the participant in collaboration with their treating pediatrician. Participants will need to inform the study team if they do not wish to be informed.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Ability to understand and follow study procedures and understand informed consent
* From week 20 of pregnancy until birth
* General good health, i.e. absence of major severe medical/ surgical/ psychiatric condition requiring ongoing management. Minor well controlled conditions (e.g. medically controlled arterial hypertension, occupational asthma, gestational diabetes mellitus) may be present.
* Absence of known severe embryonal pathology, expected normal pregnancy (e.g. minor conditions including twin/ triplet pregnancy, final pelvic position may be present)
* Age 18-45 years.

Exclusion Criteria:

• Participation in another clinical study interfering with study procedures.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: At recruitment: Healthy pregnant women in the area of Bern. On Follow-up: baby-mother pairs in the area of Bern
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-05-07 (Actual); Primary Completion 2028-03-03 (Estimated); Study Completion 2035-03-03 (Estimated)

PRIMARY OUTCOMES:
Maturation of a healthy infant intestinal microbiota regarding complexity of species composition and metabolic activities. | Infant stool samples will be collected 0-3 days after birth
  The investigators are aiming for a deep understanding of the maturation of a healthy infant intestinal microbiota considering composition, diversity and metabolic activities. The investigators will characterise the composition, metabolic potential and activity at various time points by advanced techniques (16S sequencing, metagenomics shotgun sequencing and mRNA sequencing) and the metabolites present by mass spectrometry (see "detailed description") . Using this information, the investigators will estimate networks of metabolic activity of the microbiota. Network analysis can be informed by information regarding small molecules present. The trajectories shared by the microbiota of most healthy infants will be considered normal.
Maturation of a healthy infant intestinal microbiota regarding complexity of species composition and metabolic activities. | Infant stool samples will be collected 10 days after birth
  The investigators are aiming for a deep understanding of the maturation of a healthy infant intestinal microbiota considering composition, diversity and metabolic activities. The investigators will characterise the composition, metabolic potential and activity at various time points by advanced techniques (16S sequencing, metagenomics shotgun sequencing and mRNA sequencing) and the metabolites present by mass spectrometry (see "detailed description") . Using this information, the investigators will estimate networks of metabolic activity of the microbiota. Network analysis can be informed by information regarding small molecules present. The trajectories shared by the microbiota of most healthy infants will be considered normal.
Maturation of a healthy infant intestinal microbiota regarding complexity of species composition and metabolic activities. | Infant stool samples will be collected 6 weeks after birth
  The investigators are aiming for a deep understanding of the maturation of a healthy infant intestinal microbiota considering composition, diversity and metabolic activities. The investigators will characterise the composition, metabolic potential and activity at various time points by advanced techniques (16S sequencing, metagenomics shotgun sequencing and mRNA sequencing) and the metabolites present by mass spectrometry (see "detailed description") . Using this information, the investigators will estimate networks of metabolic activity of the microbiota. Network analysis can be informed by information regarding small molecules present. The trajectories shared by the microbiota of most healthy infants will be considered normal.
Maturation of a healthy infant intestinal microbiota regarding complexity of species composition and metabolic activities. | Infant stool samples will be collected 10 weeks after birth
  The investigators are aiming for a deep understanding of the maturation of a healthy infant intestinal microbiota considering composition, diversity and metabolic activities. The investigators will characterise the composition, metabolic potential and activity at various time points by advanced techniques (16S sequencing, metagenomics shotgun sequencing and mRNA sequencing) and the metabolites present by mass spectrometry (see "detailed description") . Using this information, the investigators will estimate networks of metabolic activity of the microbiota. Network analysis can be informed by information regarding small molecules present. The trajectories shared by the microbiota of most healthy infants will be considered normal.
Maturation of a healthy infant intestinal microbiota regarding complexity of species composition and metabolic activities. | Infant stool samples will be collected 14 weeks after birth
  The investigators are aiming for a deep understanding of the maturation of a healthy infant intestinal microbiota considering composition, diversity and metabolic activities. The investigators will characterise the composition, metabolic potential and activity at various time points by advanced techniques (16S sequencing, metagenomics shotgun sequencing and mRNA sequencing) and the metabolites present by mass spectrometry (see "detailed description") . Using this information, the investigators will estimate networks of metabolic activity of the microbiota. Network analysis can be informed by information regarding small molecules present. The trajectories shared by the microbiota of most healthy infants will be considered normal.
Maturation of a healthy infant intestinal microbiota regarding complexity of species composition and metabolic activities. | Infant stool samples will be collected 24 weeks after birth
  The investigators are aiming for a deep understanding of the maturation of a healthy infant intestinal microbiota considering composition, diversity and metabolic activities. The investigators will characterise the composition, metabolic potential and activity at various time points by advanced techniques (16S sequencing, metagenomics shotgun sequencing and mRNA sequencing) and the metabolites present by mass spectrometry (see "detailed description") . Using this information, the investigators will estimate networks of metabolic activity of the microbiota. Network analysis can be informed by information regarding small molecules present. The trajectories shared by the microbiota of most healthy infants will be considered normal.
Maturation of a healthy infant intestinal microbiota regarding complexity of species composition and metabolic activities. | Infant stool samples will be collected 36 weeks after birth
  The investigators are aiming for a deep understanding of the maturation of a healthy infant intestinal microbiota considering composition, diversity and metabolic activities. The investigators will characterise the composition, metabolic potential and activity at various time points by advanced techniques (16S sequencing, metagenomics shotgun sequencing and mRNA sequencing) and the metabolites present by mass spectrometry (see "detailed description") . Using this information, the investigators will estimate networks of metabolic activity of the microbiota. Network analysis can be informed by information regarding small molecules present. The trajectories shared by the microbiota of most healthy infants will be considered normal.
Maturation of a healthy infant intestinal microbiota regarding complexity of species composition and metabolic activities. | Infant stool samples will be collected 48 weeks after birth
  The investigators are aiming for a deep understanding of the maturation of a healthy infant intestinal microbiota considering composition, diversity and metabolic activities. The investigators will characterise the composition, metabolic potential and activity at various time points by advanced techniques (16S sequencing, metagenomics shotgun sequencing and mRNA sequencing) and the metabolites present by mass spectrometry (see "detailed description") . Using this information, the investigators will estimate networks of metabolic activity of the microbiota. Network analysis can be informed by information regarding small molecules present. The trajectories shared by the microbiota of most healthy infants will be considered normal.
Maturation of a healthy infant intestinal microbiota regarding complexity of species composition and metabolic activities. | Infant stool samples will be collected 96 weeks after birth
  The investigators are aiming for a deep understanding of the maturation of a healthy infant intestinal microbiota considering composition, diversity and metabolic activities. The investigators will characterise the composition, metabolic potential and activity at various time points by advanced techniques (16S sequencing, metagenomics shotgun sequencing and mRNA sequencing) and the metabolites present by mass spectrometry (see "detailed description") . Using this information, the investigators will estimate networks of metabolic activity of the microbiota. Network analysis can be informed by information regarding small molecules present. The trajectories shared by the microbiota of most healthy infants will be considered normal.
Maturation of a healthy infant intestinal microbiota regarding complexity of species composition and metabolic activities. | Infant stool samples will be collected 5 years after birth
  The investigators are aiming for a deep understanding of the maturation of a healthy infant intestinal microbiota considering composition, diversity and metabolic activities. The investigators will characterise the composition, metabolic potential and activity at various time points by advanced techniques (16S sequencing, metagenomics shotgun sequencing and mRNA sequencing) and the metabolites present by mass spectrometry (see "detailed description") . Using this information, the investigators will estimate networks of metabolic activity of the microbiota. Network analysis can be informed by information regarding small molecules present. The trajectories shared by the microbiota of most healthy infants will be considered normal.
Maturation of a healthy infant intestinal microbiota regarding complexity of species composition and metabolic activities. | Infant stool samples will be collected 10 years after birth
  The investigators are aiming for a deep understanding of the maturation of a healthy infant intestinal microbiota considering composition, diversity and metabolic activities. The investigators will characterise the composition, metabolic potential and activity at various time points by advanced techniques (16S sequencing, metagenomics shotgun sequencing and mRNA sequencing) and the metabolites present by mass spectrometry (see "detailed description") . Using this information, the investigators will estimate networks of metabolic activity of the microbiota. Network analysis can be informed by information regarding small molecules present. The trajectories shared by the microbiota of most healthy infants will be considered normal.

SECONDARY OUTCOMES:
Impact of variations of the normal environment in Switzerland on microbiota development. | Enrolment, 0-3 days, 10 days, 6 weeks, 10 weeks, 14 weeks, 24 weeks, 36 weeks, 48 weeks, 96 weeks, 5 years and 10 years after birth.
  To understand the impact of variations of the normal environment in Switzerland on microbiota development. To this end we will use parameters for nutrition and socioeconomic status, microbiota characteristics, and metabolomics and correlate those with parameters for infant development and immunity.
Transfer of the maternal microbiota to the infant | Enrolment, 0-3 days, 10 days, 6 weeks, 10 weeks, 14 weeks, 24 weeks, 36 weeks, 48 weeks, 96 weeks, 5 years and 10 years after birth.
  To understand the transfer of the maternal microbiota to the infant. The investigators will identify bacterial species (or operational taxonomic units, OTU) in the maternal microbiota in maternal stool, maternal skin, vaginal environment, maternal placenta, as well as maternal milk at various points in time and correlate these parameters to identified species/ OTU in the intestinal and skin microbiota of the infant at various points in time (for methodology see "detailed description").
  Biological samples will be collected at:
  * Maternal vaginal swab: Enrolment.
  * Placenta swab: Birth.
  * Maternal stool and skin swabs: Enrolment, 10 days, 6 months and 1 year after birth.
  * Maternal milk samples, if nursing: 0-3 days, 10 days, 6 weeks, 10 weeks, 14 weeks, 24 weeks, 36 weeks, 48 weeks, 96 weeks after birth.
  * Infant stool and skin probes: 0-3 days, 10 days, 6 weeks, 10 weeks, 14 weeks, 24 weeks, 36 weeks, 48 weeks, 96 weeks, 5 years and 10 years after birth.
Impact of the microbiota on child development and health. | Enrolment, 0-3 days, 10 days, 6 weeks, 10 weeks, 14 weeks, 24 weeks, 36 weeks, 48 weeks, 96 weeks, 5 years and 10 years after birth.
  To understand the impact of the microbiota on child development and health. The investigators will correlate infant microbiota characteristics from the primary endpoint with
  1. Parameters for physical development (size, weight, percentiles, head circumference, mid upper arm circumference, waist to hip ratio)
  2. Parameters for neurodevelopment and child behaviour
  3. Onset/ occurrence of pathology (obesity, abdominal pain, new onset of allergies, asthma, eczema, number of infectious complications, physician consultations outside regular preventive medical checkups).
  Using questionnaires, the investigators will assess clinical parameters and parameters for child development but also acquire information regarding infectious complications, allergies and abdominal pain at enrolment and on the same follow-up dates as stated in the primary outcome section.
Impact of low resources with poor nutrition and poor hygiene in developing countries on the maturation of the intestinal microbiota | 0-3 days, 10 days, 6 weeks, 10 weeks, 14 weeks, 24 weeks, 36 weeks, 48 weeks, 96 weeks, 5 years and 10 years after birth.
  To understand the impact of low resources with poor nutrition and poor hygiene in developing countries on the maturation of the intestinal microbiota. Children from the University of Zimbabwe birth cohort were followed in a similar manner as planned for the children from the Bern infant microbiota study with the same acquisition of biological samples. The investigators will use microbiota characteristics from endpoint 1 to compare microbiota maturation in healthy Swiss infants to microbiota maturation in healthy Zimbabwean children as well as children with environmental enteropathy and stunted growth.
Effects of maternal microbiota on immunomodulatory properties of breast milk and immune maturation in the newborn | Enrolment, 0-3 days, 10 days, 6 weeks, 10 weeks, 14 weeks, 24 weeks, 36 weeks, 48 weeks, 96 weeks, 5 years and 10 years after birth.
  5) To understand the extent to which the maternal microbiota and maternal diet affects the immunomodulatory properties of breast milk and how those properties in turn influence immune maturation in the newborn, we will analyse the composition of stool and breast milk samples in regard to metabolites, cellular components, cytokines and miRNA. We will further use the material to test the impact of maternal milk in vitro (cell culture) and in vivo (mice). Immunomodulatory mechanisms will be identified and correlating changes in development and maturation of the immune system of the newborn will be analysed. (For methodology see " detailed description")

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Misselwitz, Professor, Principal Investigator — University Hospital of Bern - Insel Spital
Locations (1):
- University Hospital of Bern - Insel Spital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Participant level-data and statistical code will be published together with the results of our analyses. However, some restrictions regarding sharing of individual participant data apply according to Swiss law.

REFERENCES:
- [Derived] Cecchini L, Barmaz C, Cea MJC, Baeschlin H, Etter J, Netzer S, Bregy L, Marchukov D, Trigo NF, Meier R, Hirschi J, Wyss J, Wick A, Zingg J, Christensen S, Radan AP, Etter A, Muller M, Kaess M, Surbek D, Yilmaz B, Macpherson AJ, Sokollik C, Misselwitz B, Ganal-Vonarburg SC. The Bern Birth Cohort (BeBiCo) to study the development of the infant intestinal microbiota in a high-resource setting in Switzerland: rationale, design, and methods. BMC Pediatr. 2023 Nov 10;23(1):560. doi: 10.1186/s12887-023-04198-5. PMID 37946167

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT04447742/Prot_SAP_002.pdf
  • Informed Consent Form (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT04447742/ICF_003.pdf